CLINICAL TRIAL: NCT03825198
Title: A Prospective Randomized Double Blind Trial of the Efficacy of a Bilateral Lumbar Erector Spinae Block on the 24h Morphine Consumption After Posterior Lumbar Interbody Fusion Surgery.
Brief Title: Lumbar Erector Spinae Plane Block for Back Surgery
Acronym: LUMBES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr M. B. Breebaart (Other)
Responsible Party: Sponsor-Investigator, Dr M. B. Breebaart, senior member of staff anesthesiology department, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B300201837508
Record Dates: First submitted 2018-11-13; First posted 2019-01-31 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative; Anaesthesia; Surgery; Nerve Block; Anesthesia, Local; Back Pain; Spinal Fusion
MeSH Terms: conditions — Pain, Postoperative; Back Pain | interventions — Levobupivacaine; Sufentanil; Propofol; Rocuronium; Sevoflurane; Acetaminophen; Ketorolac; Analgesia, Patient-Controlled; Dexamethasone; Calcium Dobesilate; Morphine

STUDY DESIGN:
Intervention Model Description: double blind randomised
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The medication for the sham block with NaCl or the local anaesthetic will be prepared by an independent medical caregiver who has no connection with the patient. The anaesthetics performing the block, the patient and the observation nurses/doctors collecting the data are masked. The solutions used are not distinguishable from each other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESB group (Active Comparator): Erector Spinae plane block with 20 ml levobupivacaine 0,25% on each side. General anesthesia with 15 mcg sufentanil, 2-3 mg/kg propofol and 0,5 mg/kg Rocuronium Bromide during spine fusion surgery (1 or two intervertebral levels). Maintainance of general anesthesia with sevoflurane.
  Postoperative analgesia with Ketorolac (0,5 mg/kg), paracetamol 1000 mg (4 times/ day) and Morphine PCA. Dexamethasone is administered for the prevention of nausea.
  Interventions: Procedure: Erector spinae plane block; Drug: Levobupivacaine 0,25%; Procedure: spine fusion; Drug: Sufentanil; Drug: propofol; Drug: Rocuronium Bromide; Drug: sevoflurane; Drug: paracetamol; Drug: Ketorolac; Drug: morphine pca; Drug: Dexamethasone; Drug: Morphine
- SHAM group (Sham Comparator): Erector Spinae plane block with 20 ml NaCl 0,9% on each side General anesthesia with 15 mcg sufentanil, 2-3 mg/kg propofol and 0,5 mg/kg Rocuronium Bromide during spine fusion surgery (1 or two intervertebral levels). Maintainance of general anesthesia with sevoflurane.Postoperative analgesia with Ketorolac (0,5 mg/kg, paracetamol 1000 mg 4times/ day and Morphne PCA .Dexamethasone is administered for the prevention of nausea.
  Interventions: Procedure: Erector spinae plane block; Procedure: spine fusion; Drug: NaCL 0,9%; Drug: Sufentanil; Drug: propofol; Drug: Rocuronium Bromide; Drug: sevoflurane; Drug: paracetamol; Drug: Ketorolac; Drug: morphine pca; Drug: Dexamethasone; Drug: Morphine

INTERVENTIONS:
Procedure: Erector spinae plane block — Ultrasound guided deposition infiltration between a lumbar transverse proces and the erector spine muscle
  Other Names: Locoregional anaesthesia
Drug: Levobupivacaine 0,25% — 20 ml levobupivacaine 0,25% used for the infiltration between the transverse process and the erector spinal muscle
  Other Names: chirocaine
  Arms: ESB group
Procedure: spine fusion — fusion of lumbar vertebral body on 1 or two levels
Drug: NaCL 0,9% — 20 ml solution used for the infiltration between the transverse process and th erector spinal muscle
  Arms: SHAM group
Drug: Sufentanil — opioid used for the preoperative analgesia for back surgery during general anaesthesia ( 15 mag)
  Other Names: sufenta
Drug: propofol — induction agent for general anaesthesia ( 2-3 mg/kg)
Drug: Rocuronium Bromide — muscle relaxant used during general anaesthesia ( 0,5 mg/kg)
  Other Names: sermon
Drug: sevoflurane — inhalation aesthetic used for the maintenance of general anaesthesia
Drug: paracetamol — postoperative drug for analgesia ( 1 gram 4/day)
Drug: Ketorolac — non steroidal into inflammation drug used for postoperative analgesia (0,5 mg/kg)
Drug: morphine pca — postoperative morphine pomp, controlled by the patient. ( bolus 1 mg, lockout 8 minutes) the solution contains morphine 1 mg/ml + dehydrobenzperidol 0,05 mg/ml
  Other Names: patient controlled analgesia
Drug: Dexamethasone — drug given during general anaesthesia to prevent postoperative nausea
  Other Names: aacidexam
Drug: Morphine — loading dose morhine 0,1 mg/kg at the end of surgery

SUMMARY:
Title:

A prospective randomized double blind trial of the efficacy of a bilateral lumbar erector spinae block on the 24 h morphine consumption after posterior lumbar interbody fusion surgery.

Objectives:

The primary objective is to study the influence of a bilateral erector spinae block on 24h morphine consumption.

Endpoint:

The primary endpoint is the 24 h morphine consumption in mg. Secondary endpoints are intraoperative sufentanil requirement, total morphine during first 72 postoperative hours, NRS pain scores in rest and defined movement (moving to chair) at regular time intervals and Quality of Recovery 40 score (QoR-40) at fixed time intervals day 1 and 3 postoperatively

Population:

Patients undergoing posterior lumbar interbody fusion ranging 1 - 3 levels Phase 3

Number of sites Enrolling participants:

University Hospital Antwerp &AZ KLINA Brasschaat

Description of study agent:

Bilateral erector spinae block: each block contains 20 ml levobupivacaine 0.25% + 5 mcg/ml epinephrine Study duration Until the required study population is met Participant duration 72 hours

DETAILED DESCRIPTION:
In this prospective randomized double blind placebo controlled clinical trial we would like to assess the efficacy of a bilateral lumbar erector spinae block on the 24h morphine consumption after posterior lumbar interbody fusion surgery. Patients scheduled for 1-2 level PLIF surgery will be recruited in AZ KLINA in Brasschaat and the University Hospital Antwerp in Edegem. The study contains two arms. Subjects will be randomly allocated to an erector spinae block group or the sham block group (placebo).

Stratified randomization will be done according to gender, levels of surgery and site online with Q minim.The study medication will be prepared in identical premade syringes and numbered according to a computer generated block randomization list (1:1 ratio ESB:sham). Subjects will be assigned consecutive numbers upon inclusion to the study and receive the study medication from the corresponding numbered syringes. The study medication in syringes for injection will be prepared by an anesthesiologist neither involved in the study nor in the care of the patient, before handing it over to the investigators. The ESB-group will receive 20 ml Chirocaine 0,25%. The sham block group medication will receive 20 ml Nacl0,9%. The levobupivacaine and saline 0.9% are identical in appearance. All investigators, staff and patients will be blinded to the treatment groups. Epinephrine is added to the placebo block in order to prevent unblinding by increased heart rate or blood pressure. Unmasking will not occur until statistical analysis is complete.

Patients in the erector spinae block group will receive a bilateral ESB block with an injectate containing 20 ml of levobupivacaine 0.25% in each puncture. Patients allocated to the sham group receive a bilateral ESB block with each injectate containing 20 mL of NaCl 0.9% . The blocks will be performed by experts in the field of ultrasound guided locoregional anaesthesia namely dr D. van Aken, dr L. Sermeus and dr M.B. Breebaart who are also teachers for the BARA (Belgian Association of Regional Anaesthesia). The blocks will be performed preoperatively in a separate block room with ultrasound after placement of an iv line and application of standard monitoring (ECG, NIBP, saturation). The blocks will be placed as described by Chin et al. modified for lumbar level.8 First, the patient will be placed in the lateral or sitting position. A curve array probe or a high frequency linear probe, depending on the BMI of the patient, will be placed in a longitudinal position 2-3 cm lateral of the vertebral column. The transverse processes of the vertebrae at the (mid) level of surgery, the erector spinae muscle and the psoas muscle are identified. In case of two level surgery the transverse process of the upper level will be considered as the preferred target. Depending on the depth a 5 or 8 cm 22 G ultrasound needle (Pajunk) will be inserted with an in plane technique in a cephalad to caudad direction until bone contact with the top of the transverse process is reached. After slight retraction of the needle, 20 ml of the study medication will be injected behind the erector spinae muscle. The same procedure will be repeated on the contralateral side.

General anesthesia will then be induced in a standardized way with propofol 2-3mg/kg, sufentanil 15mcg and rocuronium 0.5mg/kg. After tracheal intubation anesthesia will be maintained with sevoflurane and intraoperative analgesia with sufentanil. The dosages of these agents will be determined at the discretion of the anesthesiologist. At the end of surgery patients will receive acetaminophen 1g IV, ketorolac (Taradyl, CSP Benelux) 0.5 mg/kg (max. 30 mg) IV and a morphine loading dose (0.1 mg/kg) IV to manage postoperative pain. Patients will be extubated in the operating theatre and admitted to the post anesthesia care unit (PACU). Postoperative pain in the PACU and on the ward will be treated with acetaminophen 1g IV round the clock (4 times daily) and by a patient controlled intravenous analgesia pump (PCIA) with morphine at a concentration of 1 mg/ml and dehydrobenzperidol (DHBP) 0.05 mg/ml. The PCIA will be set using a standardised protocol: no background administration of morphine, a bolus dose of 1.5 mL morphine with a lock-out interval of 8 minutes and an hourly limit of 7.5 mg. If pain management on the PACU is inadequate (NRS > 3) additional boli of 1 mg morphine IV will be administered with the total additional dose of morphine limited to 0.15mg/kg morphine. In case NRS is still > 3 an IV ketamine (Ketalar, Pfizer) bolus (0.2 mg/kg) will be given. All patients receive dexamethasone 5mg IV as postoperative nausea and vomiting (PONV) prophylaxis. If needed, this will be supplemented by ondansetron 4mg IV and if still insufficient with alizapride 50mg IV. Other study endpoints will be retrieved from the patient data management systems

The morphine consumption during the first 24 hours postoperatively will be extracted out of the PCIA pump. The total morphine dose requirement during the first 72 postoperative hours will also be extracted out of the PCIA pump. Pain scores at rest will be assessed with the numeric rating scale (NRS, 0=no pain 10= worst imaginable pain) and tested at regular time intervals: at the time of inclusion, at the PACU (T0 = arrival at Post Anesthesia Care Unit, T+15min, T+30min) and ward (twice daily- morning and evening until postoperative day 3) Pain scores during defined movement (first moving to chair and upright sitting) will be examined. Time to first mobilization in chair (in hours since T0) and time to first walk of twenty meters (in hours since T0) will be noted in the patients study diary. The quality of recovery 40 score (QoR-40) will be calculated out of a series of questions patients are required to answer at day 1 and 3 postoperatively. The QoR-40 is a widely used and extensively validated measure of quality of recovery. It is a 40-item questionnaire on quality of recovery from anesthesia, that has been shown to measure health status after surgery.

ELIGIBILITY:
Inclusion Criteria:

* - Patients scheduled for 1-2 level posterior lumbar interfusion surgery in AZ KLINA Hospital or University of Antwerp Hospital (UZA) after approval of Ethical Committee until all required patients are included
* American Society of Anesthesiologist (ASA) score of 1 - 3
* Age 18 - 75 year
* Normal liver and renal function

Exclusion Criteria:

* Age <18 years or mentally incompetent
* BMI < 16 or BMI > 35
* Allergy to one or more substances of the study medication (= levobupivacaine, dexamethasone, propofol, sufentanil, rocuronium, ketorolac, morphine, ketamine, DHBP, ondansetron, alizapride)
* Chronic strong opioid use (>3 intakes per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
24 hour morphine consumption | 24 hours
  total milligrams (0-150) of morphine used in the first 24 hours after surgery, extracted out of the pca pump data.

SECONDARY OUTCOMES:
Intraoperative sufentanyl requirement ( | 2-5 hours
  total Intravenous administered sufentanyl in micrograms during surgery(10-100)
Morphine consumption 72 hours | 72 hours
  total milligrams of morphine used in 72 hours after surgery (0-450), extracted out of the pca pump data
NRS pain scores | at regular intervals and defined movement until 72 hours after surgery
  Numeric rating scale pain score (in numbers) and rest (0= no pain10 =worst thinkable pain)
Quality of recovery score (QoR-40) | day 1 and day 3 postoperatively
  score in numbers of mental and psychological well being scored by list of questions (minimal score 20-maximum score 200). A high score indicates a better/faster recovery, and is inversely correlated with hospital stay
time to mobilisation to chair | 8-72 hours
  movements (mobilisation to chair) in hours after surgery
time to 20 meter walking | 8-72 hours
  movement 20 meter walking in hours after surgery

OTHER OUTCOMES:
expected preoperative pain score (NRs° | before surgery ( moment of inclusion)
  Numeric rating scale pain score (in numbers). pain that people expect before they have surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ KLina, Brasschaat, Antwerp
  - University Hospital Antwerp, Antwerp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breebaart MB, Van Aken D, De Fre O, Sermeus L, Kamerling N, de Jong L, Michielsen J, Roelant E, Saldien V, Versyck B. A prospective randomized double-blind trial of the efficacy of a bilateral lumbar erector spinae block on the 24h morphine consumption after posterior lumbar inter-body fusion surgery. Trials. 2019 Jul 17;20(1):441. doi: 10.1186/s13063-019-3541-y. PMID 31315670